CLINICAL TRIAL: NCT03996668
Title: The Effect of Compression Stockings on Cerebral Desaturation Events in Obese Patients Undergoing Shoulder Arthroscopy in the Beach Chair Position - A Randomized Prospective Study
Brief Title: Effect of Compression Stockings on Cerebral Desaturation Events in Obese Patients Undergoing Shoulder Arthroscopy in the Beach Chair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Nickolas Garbis, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 209868
Record Dates: First submitted 2019-06-11; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Shoulder Arthoscopy; Beach Chair Position; Cerebral Desaturation Events; Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients are not made aware of their study group or the presence of intraoperative cerebral desaturation events
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Subjects received standard operating room dress including sequential compression devices.
- Experimental (Experimental): Subjects wore thigh high compression stockings in addition to standard operating room dress including sequential compression devices.
  Interventions: Other: Thigh High Compression Stockings

INTERVENTIONS:
Other: Thigh High Compression Stockings — Thigh high compression stockings will be placed after induction of anesthesia and intubation.
  Arms: Experimental

SUMMARY:
The study compares the effect of thigh high compression stockings on cerebral desaturation events in patients undergoing shoulder arthroscopy in the beach chair position with a BMI greater than or equal to 30.

DETAILED DESCRIPTION:
On the day of surgery, enrolled patients whom have signed consent for participation in the study will be randomized to receive thigh high compression stockings with SCDs or SCDs alone. The importance of the investigation, proposed methodology, and potential risks of participation will be addressed. In the pre-operative holding area, a cerebral oximeter (INVOS 5100C, Covidien) will be placed on the skull as directed by the manufacturer. The sensors will be placed on the skull bilaterally in order to assess perfusion in both hemispheres. Cerebral oximeter is a non-invasive, transcutaneous tool that can be used to measure cerebral tissue oxygenation. The tool uses nearinfrared spectroscopy to measure the percentage of hemoglobin saturated with oxygen in the microcirculation of tissue within approximately 2-3cm below the skin. The technology is approved by the FDA in the anesthesia setting to monitor cerebral oxygenation and is commonly used in cardiothoracic surgery and its use has been validated in the surgical setting.11 A baseline cerebral tissue oxygen saturation (rSO2) will be recorded. All patients will be anesthetized using a standardized protocol. Once anesthesia has been induced, thigh high compression stockings will be applied to the appropriate group followed by SCDs. All patients in the study will wear sequential compression devices on both legs for thrombosis prophylaxis regardless of randomization. The patient will then be raised into the beach chair position and secured in the normal fashion and the planned surgery will begin. Intraoperative rSO2 data will be continuously recorded throughout the case. The system will be set to alarm when the rSO2 decreases greater than 20% from baseline. These events will be recorded throughout the case as CDEs. To avoid cerebral vascular injury, these events will be treated with a protocol by anesthesia including ephedrine, phenylephrine, and the patient may be returned to the supine position if needed. When surgery is complete, patients will be recovered in the post-anesthesia care unit. The study will be conducted at three facilities within the Loyola system: the Loyola Ambulatory Surgery Center at Oakbrook (LASCO), the Ambulatory Surgery Center at Loyola (ASC), and at Gottlieb Memorial Hospital (GMH). Personnel will include the attending surgeon, orthopaedic surgery residents, and anesthesia staff assigned to each case, all of whom will be fully educated on the study and protocols.

ELIGIBILITY:
Inclusion Criteria:

* • All patient over age 18

  * BMI > 30
  * Undergoing shoulder arthroscopy in beach chair position

Exclusion Criteria:

* • Age < 18 years

  * BMI < 30
  * Known and documented >90% occlusion of carotid artery
  * Prior neck surgery
  * Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Cerebral Desaturation Events | Intraoperative measurement that begins the with upright positioning and ends with return to supine positioning. There are no postoperative measures.
  Intraoperative Cerebral desaturation events is defined as a decrease of 20% or more in cerebral oxygenation percentage from a preoperative supine baseline and is measured by Near Infrared Spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Nickolas Garbis, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Pohl A, Cullen DJ. Cerebral ischemia during shoulder surgery in the upright position: a case series. J Clin Anesth. 2005 Sep;17(6):463-9. doi: 10.1016/j.jclinane.2004.09.012. PMID 16171668
- [Background] Papadonikolakis A, Wiesler ER, Olympio MA, Poehling GG. Avoiding catastrophic complications of stroke and death related to shoulder surgery in the sitting position. Arthroscopy. 2008 Apr;24(4):481-2. doi: 10.1016/j.arthro.2008.02.005. PMID 18375282
- [Background] Fischer GW, Torrillo TM, Weiner MM, Rosenblatt MA. The use of cerebral oximetry as a monitor of the adequacy of cerebral perfusion in a patient undergoing shoulder surgery in the beach chair position. Pain Pract. 2009 Jul-Aug;9(4):304-7. doi: 10.1111/j.1533-2500.2009.00282.x. Epub 2009 Mar 17. PMID 19490464
- [Background] Salazar D, Sears BW, Aghdasi B, Only A, Francois A, Tonino P, Marra G. Cerebral desaturation events during shoulder arthroscopy in the beach chair position: patient risk factors and neurocognitive effects. J Shoulder Elbow Surg. 2013 Sep;22(9):1228-35. doi: 10.1016/j.jse.2012.12.036. Epub 2013 Feb 15. PMID 23415820
- [Background] Kwak HJ, Lee JS, Lee DC, Kim HS, Kim JY. The effect of a sequential compression device on hemodynamics in arthroscopic shoulder surgery using beach-chair position. Arthroscopy. 2010 Jun;26(6):729-33. doi: 10.1016/j.arthro.2009.10.001. Epub 2010 Mar 3. PMID 20511029